CLINICAL TRIAL: NCT04653142
Title: An Open Label, Phase I Study of BI 765063 Monotherapy, and Its Combination Therapy With BI 754091, to Characterize Safety, Pharmacokinetics, and Pharmacodynamics in Japanese Patients With Advanced Solid Tumors
Brief Title: A Study to Test Different Doses of BI 765063 Alone and in Combination With BI 754091 in Japanese Patients With Different Types of Advanced Cancer (Solid Tumors)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1443-0004
Record Dates: First submitted 2020-11-27; First posted 2020-12-04 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Solid Tumors

STUDY DESIGN:
Intervention Model Description: After the completion of dose escalation with BI 765063 in Part A, Part B will commence and successive dose groups of patients will receive escalating doses of BI 765063 in combination with a fixed dose of BI 754091.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BI 765063 (Part A) and BI 765063 + BI 754091 (Part B) (Experimental)
  Interventions: Drug: BI 765063; Drug: BI 754091

INTERVENTIONS:
Drug: BI 765063 — BI 765063
Drug: BI 754091 — BI 754091

SUMMARY:
This study is open to Japanese adults with advanced cancer (solid tumors). This is a study in people for whom previous treatment was not successful and for whom no standard therapy exists. The purpose of this study is to find the highest dose of BI 765063 that people can tolerate when taken alone or together with a medicine called BI 754091. BI 765063 and BI 754091 are antibodies that may help the immune system fight cancer (checkpoint inhibitors).

Participants get BI 765063 alone or together with BI 754091 as infusion every 3 weeks.

Participants can stay in the study as long as they benefit from treatment and can tolerate it. The doctors check the health of the participants and note any health problems that could have been caused by BI 765063 or BI 754091.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated the written informed consent form (ICF) prior to any trial-specific procedures
2. Male or female aged ≥ 20 years (no upper limit of age) at the time of ICF signature
3. Patients who were born in Japan, and have lived outside Japan <10 years
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at the screening visit
5. Life expectancy of at least 3 months
6. Patients with at least one Signal Regulatory Protein-alpha (SIRPα) V1 allele will be selected, i.e. homozygous V1/V1 or heterozygous V1/V2; SIRPα polymorphism will be assessed in blood sampling (patient DNA); V1 allele is understood to include V1 and V1-like alleles
7. Patients with histologically or cytologically documented advanced/metastatic primary or recurrent solid tumors who failed or are not eligible to standard therapy
8. Patients with at least one measurable lesion as per RECIST v1.1 Further inclusion criteria apply.

Exclusion Criteria:

1. Patients without at least one SIRPα V1 allele, i.e. SIRPα V2/V2 individuals
2. Previous treatment with study medications in this trial
3. Patients with symptomatic/active central nervous system (CNS) metastases. Patients with previously treated brain metastases are eligible, if there is no evidence of progression for at least 28 days before the first study drug administration without requirement for treatment with corticosteroids, as ascertained by clinical examination and brain imaging magnetic resonance imaging (MRI) or computed tomography (CT)) during the screening period
4. Any tumor location necessitating an urgent therapeutic intervention (e.g., palliative care, surgery or radiation therapy, such as spinal cord compression, other compressive mass, uncontrolled painful lesion, bone fracture)
5. Presence of active invasive cancers other than the one treated in this trial within 5 years prior to screening, except appropriately treated basal cell carcinoma of the skin, or in situ carcinoma of uterine cervix, or other local tumors considered cured by local treatment
6. Patients with active autoimmune disease or a documented history of autoimmune disease, that requires systemic treatment, i.e. corticosteroids or immunosuppressive drugs, except patients with vitiligo, resolved childhood asthma/atopy, alopecia, or any chronic skin condition that does not require systemic therapy, patients with autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone and/or controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible
7. Patients who has experienced severe infusion related reaction (IRR) to monoclonal antibody (mAb) (Grade ≥ 3 NCI CTCAE v5.0)
8. Patients removed from previous anti-PD-1 or anti-PD-L1 therapy because of a severe, or life-threatening immune related adverse event (irAE) (Grade ≥ 3 NCI CTCAE v5.0) Further exclusion criteria apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of BI 765063, Part A | up to 3 weeks
Maximum Tolerated Dose (MTD) of BI 765063, Part B | up to 3 weeks
Number of patients with dose limiting toxicity (DLT) in the MTD evaluation period, Part A | up to 3 weeks
Number of patients with dose limiting toxicity (DLT) in the MTD evaluation period, Part B | up to 3 weeks

SECONDARY OUTCOMES:
Number of patients with DLTs, Part A | 3 weeks per treatment cycle
Number of patients with DLTs, Part B | 3 weeks per treatment cycle
Percentage of patients with drug related Adverse Events (AE), Part A | 3 weeks per treatment cycle
Percentage of patients with drug related Adverse Events (AE), Part B | 3 weeks per treatment cycle
Cmax (maximum concentration) for BI 765063, Part A | up to 3 weeks
Cmax (maximum concentration) for BI 765063, Part B | up to 3 weeks
Cmax (maximum concentration) for BI 754091, Part B | up to 3 weeks
AUC0-tz (area under the curve) for BI 765063, Part A | up to 3 weeks
AUC0-tz (area under the curve) for BI 765063, Part B | up to 3 weeks
AUC0-tz (area under the curve) for BI 754091, Part B | up to 3 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- Japan (4):
  - National Cancer Center Hospital East, Chiba, Kashiwa
  - Shikoku Cancer Center, Ehime, Matsuyama
  - Osaka International Cancer Institute, Osaka, Osaka
  - National Cancer Center Hospital, Tokyo, Chuo-ku

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com/